CLINICAL TRIAL: NCT03251547
Title: Recombinant Activated Factor VII (rFVIIa/ NovoSeven®) in the Management of Massive Bleeding in Hospital Universiti Sains Malaysia
Brief Title: Recombinant Activated Factor VII in the Management of Massive Bleeding in Hospital Universiti Sains Malaysia
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Soon Eu Chong, Dr, Universiti Sains Malaysia
Other Study IDs: SEChong
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Massive Hemorrhage; Massive Blood Loss; Massive Blood Transfusion; Thrombocytopenia
Keywords: rFVIIa; Massive Hemorrhage; non-hemophilia
MeSH Terms: conditions — Thrombocytopenia | interventions — recombinant FVIIa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NovoSeven: Non-hemophiliac patients experienced massive haemorrhage who was treated with recombinant activated factor VII
  Interventions: Drug: NovoSeven

INTERVENTIONS:
Drug: NovoSeven — To survey retrospectively the treatment indications, clinical outcome, transfusion need and changes in coagulation profiles of non-haemophiliac patients who had received rFVIIa during massive bleeding
  Other Names: recombinant activated factor VII

SUMMARY:
This is a retrospective descriptive study, to study the treatment indications, changes in transfusion need, coagulation profiles changes and clinical outcome (survival, complication) of non-haemophiliac patients who received activated factor seven (rFVIIa / NovoSeven®) during massive bleeding in Hospital Universiti Sains Malaysia (HUSM)

DETAILED DESCRIPTION:
Effective hemostasis can be life-saving. However, there is still lack of an ideal hemostatic drug which is safe and effective.

Recombinant activated factor VII (rFVIIa; Novo Nordisk, Bagsvaerd, Denmark) is a hemostatic agent originally developed for the management of bleeding in haemophilia A and B patients with inhibitors to factor VIII or IX respectively.

Recombinant FVIIa involves in extrinsic clotting pathway where it forms a complex with tissue factor which in the presence of calcium and phospholipids activates coagulation factor X which then initiates the conversion of prothrombin into thrombin at the site of injury (Figure 1). Formation of thrombin and clot stabilises platelet plug and form a tight fibrin structure which is resistant to lysis. Due to the efficient haemostatic property but the unknown safety profile, it is only being used as one of the last resorts during massive intractable bleeding episode among the non-haemophilia patients.

Efficacy and safety profile is the most important concern of a haemostatic drug like rFVIIa. However, there is ongoing controversial evidence regarding thromboembolic complications and survival benefit of the off-label use of rFVIIa in massive bleeding (Patel et al2012).

This a study to learn about the previous usage, outcome and complications of rFVIIa use in massive intractable bleeding management in a single centre (Hospital University Sains Malaysia / HUSM) in Malaysia.

The data of patients who had undergone massive bleeding will be available from pharmacy department and recruited from medical record department of HUSM.

These include:

1. Underlying condition, BMI of patient.
2. Indication for blood transfusion.
3. Dose of rFVIIa.
4. Other medication (vitamin K, tranexamic acid, anticoagulant, antiplatelet) given to patient.
5. Blood pressure, haemoglobin level, coagulation profile, and blood product requirements 24 hours before and after administration of rFVIIa.
6. Survival at 24-hour and day-30 post administration of rFVIIa were also recorded.
7. Thromboembolism complication post administration of rFVIIa.
8. Duration of stay.

Patients' identities will be anonymized without disclosure of personal identifiable information to third-party organizations.

Statistical calculations will be done using SPSS (Statistical Package for the Social Science) software.

Quantitative data will be expressed as mean ± standard deviation (SD) and median (interquartile range,IQR). For comparison before and after of administration of rFVIIa, data will be analyzed using paired t- test if the data is normally distributed. For skewed data, Wilcoxon Signed-Rank test will be used for analysis. The differences willl be considered significant at a p < 0.05.

For the outcome of survival and thromboembolic complication, data will be analyzed descriptively with frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* All patient with massive bleeding who had received rFVIIa from year 2006 to year 2016.
* Massive bleeding criteria

  * Loss of one blood volume within a 24 hour
  * 50% blood volume loss within 3 h
  * Rate of loss of 150 ml/min

Exclusion Criteria:

* Haemophilia patient who received rFVIIa
* Poor documentation / record unavailable in HUSM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-haemophilic patients who had received rFVIIa during massive bleeding in Hospital Universiti Sains Malaysia (HUSM)
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in blood transfusion requirement | 24 hour before and after administration of rFVIIa
  To study the changes in blood product requirement in 24 hours before and after administration of rFVIIa in massive bleeding patient in HUSM and to describe the factors affecting it.
Survival rate | 30 days
  To describe the outcome of survival at 24-hour and Day-30 after receiving rFVIIa

SECONDARY OUTCOMES:
Changes in coagulation profile | 24 hour before and after administration of rFVIIa
  To study the changes in coagulation profile in 24 hours before and after administration of rFVIIa in massive bleeding patient in HUSM and to describe the factors affecting it

OTHER OUTCOMES:
Complication rate | 30 days
  To describe the outcome of complication of non-hemophiliac patient after receiving rFVIIa

CONTACTS AND LOCATIONS:
Overall Officials: Chong Soon Eu, MD, MMed, Study Chair — Universiti Sains Malaysia; Nurfatin Mohd Shah, BSc, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hunt BJ. Bleeding and coagulopathies in critical care. N Engl J Med. 2014 Feb 27;370(9):847-59. doi: 10.1056/NEJMra1208626. No abstract available. PMID 24571757
- [Background] Bougle A, Harrois A, Duranteau J. Resuscitative strategies in traumatic hemorrhagic shock. Ann Intensive Care. 2013 Jan 12;3(1):1. doi: 10.1186/2110-5820-3-1. PMID 23311726
- [Background] Cosgriff N, Moore EE, Sauaia A, Kenny-Moynihan M, Burch JM, Galloway B. Predicting life-threatening coagulopathy in the massively transfused trauma patient: hypothermia and acidoses revisited. J Trauma. 1997 May;42(5):857-61; discussion 861-2. doi: 10.1097/00005373-199705000-00016. PMID 9191667
- [Background] Faraoni D, Van Der Linden P. A systematic review of antifibrinolytics and massive injury. Minerva Anestesiol. 2014 Oct;80(10):1115-22. Epub 2013 Nov 28. PMID 24287671
- [Background] Franchini M. The use of desmopressin as a hemostatic agent: a concise review. Am J Hematol. 2007 Aug;82(8):731-5. doi: 10.1002/ajh.20940. PMID 17492648
- [Background] Kobayashi T, Nakabayashi M, Yoshioka A, Maeda M, Ikenoue T. Recombinant activated factor VII (rFVIIa/NovoSeven(R)) in the management of severe postpartum haemorrhage: initial report of a multicentre case series in Japan. Int J Hematol. 2012 Jan;95(1):57-63. doi: 10.1007/s12185-011-0974-9. Epub 2011 Dec 9. PMID 22160834
- [Background] Lin Y, Moltzan CJ, Anderson DR; National Advisory Committee on Blood and Blood Products. The evidence for the use of recombinant factor VIIa in massive bleeding: revision of the transfusion policy framework. Transfus Med. 2012 Dec;22(6):383-94. doi: 10.1111/j.1365-3148.2012.01164.x. Epub 2012 May 27. PMID 22630348
- [Background] Logan AC, Goodnough LT. Recombinant factor VIIa: an assessment of evidence regarding its efficacy and safety in the off-label setting. Hematology Am Soc Hematol Educ Program. 2010;2010:153-9. doi: 10.1182/asheducation-2010.1.153. PMID 21239786
- [Background] Palmason R, Vidarsson B, Sigvaldason K, Ingimarsson JP, Gudbjartsson T, Sigurdsson GH, Onundarson PT. Recombinant factor VIIa as last-resort treatment of desperate haemorrhage. Acta Anaesthesiol Scand. 2012 May;56(5):636-44. doi: 10.1111/j.1399-6576.2012.02688.x. PMID 22489992
- [Background] Spahn DR, Bouillon B, Cerny V, Coats TJ, Duranteau J, Fernandez-Mondejar E, Filipescu D, Hunt BJ, Komadina R, Nardi G, Neugebauer E, Ozier Y, Riddez L, Schultz A, Vincent JL, Rossaint R. Management of bleeding and coagulopathy following major trauma: an updated European guideline. Crit Care. 2013 Apr 19;17(2):R76. doi: 10.1186/cc12685. PMID 23601765
- [Background] Stainsby D, MacLennan S, Hamilton PJ. Management of massive blood loss: a template guideline. Br J Anaesth. 2000 Sep;85(3):487-91. doi: 10.1093/bja/85.3.487. PMID 11103199
- [Background] Yank V, Tuohy CV, Logan AC, Bravata DM, Staudenmayer K, Eisenhut R, Sundaram V, McMahon D, Olkin I, McDonald KM, Owens DK, Stafford RS. Systematic review: benefits and harms of in-hospital use of recombinant factor VIIa for off-label indications. Ann Intern Med. 2011 Apr 19;154(8):529-40. doi: 10.7326/0003-4819-154-8-201104190-00004. PMID 21502651